CLINICAL TRIAL: NCT01559961
Title: A Phase I Dose Escalation Study of the Safety and Pharmacokinetics of Single Intravesical Doses of TTI-1612 in Women With Interstitial Cystitis/Bladder Pain Syndrome
Brief Title: Safety Study of Single Intravesical Doses of TTI-1612 in Women With Interstitial Cystitis/Bladder Pain Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trillium Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTI-IC-0111-SAD
Record Dates: First submitted 2012-03-15; First posted 2012-03-21 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Interstitial Cystitis
Keywords: bladder; cystitis; frequency; nocturia; pain; urgency
MeSH Terms: conditions — Cystitis, Interstitial; Cystitis; Nocturia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TTI-1612 (Experimental): Single intravesical 30-minute treatments with escalating doses of TTI-1612.
  Interventions: Drug: TTI-1612

INTERVENTIONS:
Drug: TTI-1612 — Single intravesical 30-minute treatments with escalating doses of TTI-1612.

SUMMARY:
The purpose of this study is to determine the safety and pharmacokinetics of TTI-1612 in women with interstitial cystitis/bladder pain syndrome.

DETAILED DESCRIPTION:
Single doses of TTI-1612, at seven escalating dose levels, will be administered intravesically to women with IC/BPS. Drug will be retained in the bladder for 30 minutes.

TTI-1612 pharmacokinetics will be studied through the collection of blood samples at various time points, from 5 minutes to 8 hours post administration on dosing day, then at 24 and 48 hours post dosing. Serum will be isolated for subsequent analysis and determination of the following parameters: maximum serum concentration (Cmax), time of maximum observed concentration (Tmax), area under the curve to the final time with a concentration above the limit of quantification (AUC 0-t) and to infinity (AUC 0-∞), elimination half-life (t½), clearance (CL) and volume of distribution (Vz).

TTI-1612 safety will be determined through monitoring of the subjects' vital signs, ECGs, clinical laboratory evaluations, adverse events (if any) and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female, 18 to 65 years old, inclusive.
* Subject has read and signed an ICF.
* Subject has BMI of 18 to 32kg/sq.m., inclusive.
* Subject has been diagnosed with IC/BPS, according to current AUA guidelines for IC/BPS.
* Subjects of child-bearing potential must agree: (1) to a double-barrier contraception method between screening and baseline visits, and (2) to abstain from sexual intercourse from baseline visit through to study completion (day 7 +/- 1 day).
* Subject has a negative serum pregnancy test at screening and at baseline.
* Subject is not lactating.
* Subject has documented negative antibody tests for HIV, HbSAg or HCV within 3 months prior to dosing or tests negative at screening.
* Subject tests negative for bladder cancer by cystoscopy within 6 months prior to dosing and tests negative by urine cytology at screening.
* Subject has clinical laboratory values (CBCs, comprehensive metabolic panel and urinalysis) that fall within normal ranges or are not clinically significant in the opinion of the Investigator.

Exclusion Criteria:

* Subject has a history of oncologic disease except non-melanoma skin cancer.
* Subject has any other condition that, in the opinion of the Investigator, may jeopardize the safety of the subject or may impact the validity of the study results.
* Subject, for whatever reason, has had substantial changes in eating habits within 30 days prior to dosing, which, in the opinion of the Investigator, may confound the planned PK evaluations or interpretation of the results of the study.
* Subject has donated blood within 30 days or plasma within 14 days prior to dosing.
* Subject has used intravesical therapy within 3 months prior to dosing.
* Subject is receiving non-stable therapy for IC/BPS (stable therapy is defined as continuous treatment for at least 6 months).
* Subject has used an investigational agent within 3 months prior to dosing.
* Subject has an ECG or vital signs at baseline that, in the opinion of the Investigator or Sponsor, is/are clinically significant.
* Subject has consumed alcohol, grapefruit, grapefruit juice or xanthine-containing beverages or foods within 48 hours prior to dosing.
* Subject has taken any known hepatic enzyme-altering drugs within 30 days prior to dosing.
* Subject has taken any known heparin-containing drugs within 30 days prior to dosing.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of TTI-1612 | 7 days
  Adverse events, physical examinations, ECGs, vital signs and clinical laboratory evaluations.

SECONDARY OUTCOMES:
Pharmacokinetics | 5 minutes to 48 hours post dosing
  Blood samples will be obtained pre-dose, at 5, 10, 15, 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 24, 48 hours post dosing. Serum will be analyzed for levels of TTI-1612.
  The following parameters will be evaluated:
  * C(max) - maximum concentration,
  * T(max) - time to maximum concentration,
  * AUC(0-t) - area under the curve from time zero to the final time with a concentration above the limit of quantification,
  * AUC(0-∞) - area under the curve from time zero to infinity,
  * T(1/2) - elimination half-life,
  * CL - clearance,
  * V(z) - volume of distribution during the terminal phase.

CONTACTS AND LOCATIONS:
Overall Officials: Penka Petrova, PhD, Study Director — Trillium Therapeutics Inc.
Locations (4):
- Canada (4):
  - Bramalea Medical Centre, Brampton, Ontario
  - Urology Associates/Urologic Medical Research, Kitchener, Ontario
  - The Fe/Male Health Centres, Oakville, Ontario
  - Urology & Male Fertility Clinic, Toronto, Ontario